CLINICAL TRIAL: NCT05484557
Title: Prevention of Thromboembolism Using Apixaban vs Enoxaparin Following Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loewenstein Hospital (Other)
Responsible Party: Principal Investigator, amiram-catz, Head of the spinal department, Loewenstein Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0023-20-LOE
Record Dates: First submitted 2022-07-24; First posted 2022-08-02 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Spinal Cord Injuries; Spinal Diseases
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Diseases | interventions — apixaban; enoxaparin sodium

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study (Experimental): treatment with Apixaban
  Interventions: Drug: Apixaban
- Control (Active Comparator): treatment with Enoxaparin
  Interventions: Drug: Enoxaparin Sodium

INTERVENTIONS:
Drug: Apixaban — treatment for 6 to 12 weeks
  Arms: study
Drug: Enoxaparin Sodium — treatment for 6 to 12 weeks
  Arms: Control

SUMMARY:
Currently, Enoxaparin is the usual prophylactic anticoagulant treatment at the acute and sub-acute phases of spinal cord injury (SCI). Patients at the sub-acute phase of SCI (rehabilitation) will be given either Enoxaparin 40 mg/day (control) or Apixaban 2.5-5 mg twice a day. Apixaban dose will be determined by the treating physician. Treatment will be continued for either 6 or 12 weeks following injury (for AIS grades C-D and A-B respectively).

Endpoints: Venous thromboembolism will be evaluated by D-Dimer test every 2 weeks and an ultrasound doppler at the beginning and the end of the treatment. Bleeding events will be recorded and hematocrit will be monitored every two weeks.

ELIGIBILITY:
Inclusion Criteria:

* spinal cord injury (traumatic of not traumatic), Hebrew speaker.

Exclusion Criteria:

* contra-indication for anticoagulant treatment
* concomitant treatment with any other anticoagulant
* anticoagulant treatment needed for indications other than VTE prevention following spinal cord injury
* active clinically significant bleeding
* any lesion or condition considered a significant risk factor for major bleeding.
* hepatic disease associated with coagulopathy and clinically relevant bleeding risk
* pregnancy or breast-feeding
* heart valve related issues
* galactose intolerance
* active cancer
* patients who require thrombolysis or pulmonary embolectomy
* patients with renal impairment
* sensitivity to excipients of the medication
* anti phospholipid syndrome
* prosthetic heart valve
* acute ischemic stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants with venous thromboembolism (VTE) | 2 years
  deep vein thrombosis or pulmonary embolism

SECONDARY OUTCOMES:
Number of participants with bleeding events. | 6 to 12 weeks
  bleeding occurrence (decrease of hemoglobin by at least 1 g/dL) during the medication period.

CONTACTS AND LOCATIONS:
Locations (1):
- Loewenstein Rehabilitation Hospital, Raanana, Israel

IPD SHARING:
Plan to Share IPD: No